CLINICAL TRIAL: NCT03080701
Title: Systems of Support (SOS) to Increase Colon Cancer Screening Disparities Supplement
Brief Title: Financial Incentives to Increase Colorectal Cancer Screening in Priority Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of Michigan (Other); University of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 4RO1CA121125-09 REVISED; 4R01CA121125-09 (NIH)
Record Dates: First submitted 2017-01-31; First posted 2017-03-15 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Colorectal Cancer
Keywords: Behavioral: Automated Mailing
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The randomization sequence will be concealed to everyone except the study biostatistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - Automated Mailing (No Intervention): The mailing process will be identical to those used in the SOS study. Mailing 1 includes an introductory letter on CRC screening and a pamphlet on CRC testing choices (colonoscopy every 10 years, FIT testing yearly, or flexible sigmoidoscopy every 10 years combined with interval FIT testing), and pros and cons of each. The letter will state that they will soon be receiving a FIT kit in the mail, and a number to call if they prefer another option. Mailing 2 includes a brief letter reaffirming the importance of screening, a FIT kit (the one used by Group Health), pictograph instructions, and a postage-paid return envelope. Mailing 3 a reminder letter, is sent to participants not completing the FIT kit after 3 weeks. The intervention for Group 1 includes no incentive.
- Group 2 - Auto Mailing Plus Money (Experimental): Receives the same number of mailings and materials as group 1 with the following modifications. In Mailing 1 the letter will include the intervention notification that they will receive a monetary thank you gift for completing testing (FIT colonoscopy or flex sig within 6 months). Mailing 2 and mailing 3 (reminder letters for those still not returning kits) will include the same information about the monetary thank you gift for CRC screening completion. Mailing 4 will include the money with a thank you letter for those who complete the screening
  Interventions: Behavioral: Auto Mailing Plus Money
- Group 3 - Auto Mailing Plus Lottery (Experimental): Receives the same number of mailings and materials as group 1 with the following modifications. In Mailing 1 the letter will include the intervention notification that they will have a 1 in 10 chance of winning money (FIT, colonoscopy or flex sig within 6 months). Mailing 2 and mailing 3 (reminder letters for those still not returning kits) will include the same information about the 1 in 10 chance of winning the lottery for CRC screening completion. Mailing 4 will include a thank you letter with money for those who complete their screening and win the lottery. Participants who do not win the lottery will receive a thank you letter.
  Interventions: Behavioral: Auto Mailing Plus Lottery

INTERVENTIONS:
Behavioral: Auto Mailing Plus Money — Participant receives money as a thank you for completing CRC screening within 6 months.
  Arms: Group 2 - Auto Mailing Plus Money
Behavioral: Auto Mailing Plus Lottery — Participant has a 1 in 10 chance of winning money in a lottery for completing CRC screening within 6 months.
  Arms: Group 3 - Auto Mailing Plus Lottery

SUMMARY:
The investigators propose to build on the success of the Systems of Support to Increase Colorectal Cancer trial (SOS, R01CA121125, Green) and focus on disparity groups who are less likely to be current for colorectal cancer (CRC) screening. We will test whether financial incentives increases screening uptake and decreases screening disparities. The investigators hypothesize that CRC screening rates will be higher in patients offered mailed fecal kits and financial incentives than those offered mailed fecal kits alone.

DETAILED DESCRIPTION:
Study staff will send invitation letters and a questionnaire to 5,000 patients aged 50-75 not current for CRC screening, two-thirds who are identified in the electronic data as being from a non-White race, ethnicity, or who have Medicaid coverage. Those returning the survey and remaining eligible (estimated N = 1150) will be randomized to either (1) Mailed fecal kit only, or mailed fecal kit plus one of 2 types of financial incentives for completing testing: (2) a guaranteed Monetary incentive or (3) a probabilistic Lottery incentive.

ELIGIBILITY:
Inclusion Criteria:

* No evidence in electronic data of FIT screening in past year or a colonoscopy in the prior 9 years.
* Continuously enrolled in Group Health Cooperative (GHC) for at least one year.
* Patients who have Medicaid coverage or are non-white race or Hispanic any race.

Exclusion Criteria:

* Known high risk for CRC
* History of CRC
* History of inflammatory bowel disease
* Current anticoagulation therapy
* Organ failure
* Serious illness
* Debilitating disease
* Dementia
* Nursing home resident

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 898 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
CRC Screening Within 6 Months Following Randomization | 6 months
  We will compare among the 3 arms (1) automated mailing; (2) Auto mailing plus $10; (3) Auto mailing plus $50 lottery for completion and the effect of each on CRC screening completion at 6 months (yes/no) within the following subgroups of each arm: 1. White and not Hispanic versus non-White or Hispanic. 2. Medicaid versus non-Medicaid (Medicare, employer-based, private) insurance. 3. History of prior versus no prior completion of CRC screening tests. 4. High school or less versus college or more education level.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly B Green, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No